CLINICAL TRIAL: NCT01711658
Title: TRYHARD: A Phase II, Randomized, Double Blind, Placebo-Controlled Study of Lapatinib (Tykerb®) for Non-HPV Locally Advanced Head and Neck Cancer With Concurrent Chemoradiation
Brief Title: TRYHARD: Radiation Therapy Plus Cisplatin With or Without Lapatinib in Treating Patients With Head and Neck Cancer.
Acronym: TRYHARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RF-3501; LAP116153 (Other: GlaxoSmith Kline, LLC)
Record Dates: First submitted 2012-10-16; First posted 2012-10-22 (Estimated); Results first posted 2021-11-29 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2021-10

CONDITIONS: Non-HPV Locally Advanced Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Lapatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMRT + cisplatin + placebo (Placebo Comparator): Intensity Modulated Radiation Therapy (IMRT) with cisplatin and placebo
  Interventions: Radiation: IMRT; Drug: Cisplatin; Drug: placebo
- IMRT + cisplatin + lapatinib (Active Comparator): IMRT with cisplatin and lapatinib
  Interventions: Radiation: IMRT; Drug: Cisplatin; Drug: Lapatinib

INTERVENTIONS:
Radiation: IMRT — Intensity modulated radiation therapy (IMRT), 35 fractions over 6 weeks, 6 fractions per week for 5 weeks and 5 fractions per week for 1 week, 2 Gy per fraction to total dose of 70 Gy
Drug: Cisplatin — 100 mg/m^2 administered intravenously on days 8 and 29
Drug: placebo — 1500 mg placebo daily by mouth or by feeding tube starting 7 days before IMRT for 7 weeks prior to and during IMRT and 3 months after completion of IMRT
  Arms: IMRT + cisplatin + placebo
Drug: Lapatinib — 1500 mg lapatinib by mouth or by feeding tube daily starting 7 days before IMRT for 7 weeks prior to and during IMRT and 3 months after completion of IMRT
  Arms: IMRT + cisplatin + lapatinib

SUMMARY:
PURPOSE: This trial is studying if and how well lapatinib adds to the effectiveness of radiation therapy plus cisplatin in patients who have head and neck cancer that is not related to the human papillomavirus (HPV).

ELIGIBILITY:
Inclusion criteria:

* Patients must have histologically or cytologically confirmed diagnosis (from primary lesion and/or lymph nodes) of Squamous Cell Cancer of the oropharynx, hypopharynx or larynx (For patients with oropharynx primary, the tumor must be negative for p16 by immunohistochemistry).
* Patients with selected Stage III or IV disease (T2 N2-3 M0, T3-4 any N M0, T1 N2b, N2c or N3 p16 negative oropharynx cancer or T1-2 any N+ hypopharynx cancer) including no distant metastases.
* History/Physical examination by a Radiation Oncologist and Medical oncologist prior to entering the study.
* Examination by an ears, nose, throat (ENT) or Head & Neck Surgeon including laryngopharyngoscopy prior to entering the study.
* Patients must have a chest CT scan, or positron emission tomography (PET)/CT scan to rule out metastatic disease
* Patients must have a contrast enhanced CT scan or MRI or PET/CT scan of the tumor site and neck nodes prior to entering the study.
* Patients must have an EKG and echocardiogram (ECHO) or multigated acquisition (MUGA) scan prior to entering the study.
* Patients must have Zubrod Performance Status of 0-1.
* Patients must be ≥ 18 years of age.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 8.0 g/dl
  * Serum creatinine < 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min
  * Total bilirubin < 2 x the institutional upper limit of normal
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x the institutional upper limit of normal
* Patient must have magnesium, calcium, glucose, potassium and sodium levels within normal limits
* Women of childbearing potential must have a negative pregnancy test prior to registration.
* Patients of reproductive potential must practice effective contraception while on study and for at least 60 calendar days following treatment.
* All patients must sign an informed consent prior to enrollment.
* Patients must comply with the treatment plan and follow-up schedule.

Exclusion criteria:

* Patients with simultaneous primaries or bilateral tumors.
* Patients who have had gross total excision of the primary tumor.
* Patients with initial surgical treatment, radical or modified neck dissection.
* Patients who received prior systemic chemotherapy for the study cancer.
* Patients who received prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Patients with primary tumor of oral cavity, nasopharynx, sinuses or salivary glands.
* Prior allergic reaction to the study drugs.
* Patients who have had prior therapy that specifically and directly targets the epidermal growth factor receptor (EGFR)/human epidermal growth factor receptor 2 (HER2) pathway.
* Patients who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment);
* Pregnant women or sexually active patients not willing or able to use medically acceptable forms of contraceptive method while on treatment.
* Patients with severe, active co-morbidity, defined as follows:

  * Uncontrolled cardiac disease, such as uncontrolled hypertension, unstable angina, and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Left ventricular ejection fraction < 45%
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 calendar days prior to registration
  * Hepatic insufficiency resulting in clinical jaundice and/or Coagulation defects
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Wong, MD, Principal Investigator — Medical College of Wisconsin
Locations (16):
- United States (15):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of California, San Diego, La Jolla, California
  - Sutter General Hospital, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - University of Texas Southwestern Medical School, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- McGill Cancer Centre at McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Harrington K. et al. Phase II study of oral Lapatinib, a dual-tyrosine kinase inhibitor, combined with chemoradiotherapy (CRT) in patients with advanced squamous cell carcinoma of the head and neck (SCCHN). J Clin Oncol. 28:15s, 2010 suppl. Abstract 5505. GSK study 884
- [Derived] Wong SJ, Torres-Saavedra PA, Saba NF, Shenouda G, Bumpous JM, Wallace RE, Chung CH, El-Naggar AK, Gwede CK, Burtness B, Tennant PA, Dunlap NE, Redman R, Stokes WA, Rudra S, Mell LK, Sacco AG, Spencer SA, Nabell L, Yao M, Cury FL, Mitchell DL, Jones CU, Firat S, Contessa JN, Galloway T, Currey A, Harris J, Curran WJ Jr, Le QT. Radiotherapy Plus Cisplatin With or Without Lapatinib for Non-Human Papillomavirus Head and Neck Carcinoma: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2023 Nov 1;9(11):1565-1573. doi: 10.1001/jamaoncol.2023.3809. PMID 37768670

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After first step registration and prior to randomization, patients with oropharyngeal cancer were tested for p16. Only patients with p16-negative tumors continued to randomization. Patients with larynx or hypopharynx cancer did not require p16 testing. In total, 142 patients were enrolled and 127 were randomized.
Groups:
- IMRT + Cisplatin + Placebo: Intensity Modulated Radiation Therapy (IMRT), 35 fractions over 6 weeks, 6 fractions per week for 5 weeks and 5 fractions per week for 1 week, 2 Gy per fraction to total dose of 70 Gy
  Cisplatin: 100 mg/m^2 administered intravenously on days 8 and 29
  Placebo: 1500 mg placebo daily by mouth or by feeding tube starting 7 days before IMRT for 7 weeks prior to and during IMRT and 3 months after completion of IMRT
- IMRT + Cisplatin + Lapatinib: IMRT: IMRT, 35 fractions over 6 weeks, 6 fractions per week for 5 weeks and 5 fractions per week for 1 week, 2 Gy per fraction to total dose of 70 Gy
  Cisplatin: 100 mg/m^2 administered intravenously on days 8 and 29
  Lapatinib: 1500 mg lapatinib by mouth or by feeding tube daily starting 7 days before IMRT for 7 weeks prior to and during IMRT and 3 months after completion of IMRT
Period: Overall Study
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Started | 64 | 63
Participants Who Started Protocol Treatment | 59 | 60
Completed (Participants contributing data to results are considered to have completed the study.) | 64 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- IMRT + Cisplatin + Placebo: IMRT: IMRT, 35 fractions over 6 weeks, 6 fractions per week for 5 weeks and 5 fractions per week for 1 week, 2 Gy per fraction to total dose of 70 Gy
  Cisplatin: 100 mg/m^2 administered intravenously on days 8 and 29
  Placebo: 1500 mg placebo daily by mouth or by feeding tube starting 7 days before IMRT for 7 weeks prior to and during IMRT and 3 months after completion of IMRT
- Total: Total of all reporting groups
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Median (Full Range); unit: years] | 58 [42 to 80] | 57 [33 to 75] | 58 [33 to 80]
Age, Customized [Count of Participants; unit: Participants]
  <=65 | 54 | 56 | 110
  >65 | 10 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 51 | 47 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 60 | 61 | 121
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 9 | 10 | 19
  White | 49 | 50 | 99
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 33 | 27 | 60
    1 | 31 | 36 | 67
Smoking history: pack-years [Median (Full Range); unit: pack-years] — Smoking history as measured in pack-years. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked. Population: Two patients are missing smoking history data.
  pack-years
    number analyzed (Participants) | 63 | 62 | 125
    (all) | 38 [0 to 126] | 29.5 [0 to 168] | 30 [0 to 168]
Smoking history: pack-years [Count of Participants; unit: Participants] — Smoking history as measured in pack-years. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked. Population: Two patients are missing smoking history data.
  Participants
    number analyzed (Participants) | 63 | 62 | 125
    <=10 | 13 | 17 | 30
    >10 | 50 | 45 | 95
Primary site [Count of Participants; unit: Participants] — Primary location of tumor.
  Participants
    Oropharynx, p16-negative (central review) | 15 | 16 | 31
    Oropharynx, unknown p16 (central review) | 0 | 1 | 1
    Hypopharynx | 16 | 7 | 23
    Larynx | 33 | 39 | 72
T stage (stratification factor) [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    T1 | 2 | 0 | 2
    T2 | 9 | 7 | 16
    T3 | 35 | 38 | 73
    T4 | 18 | 18 | 36
N stage (stratification factor) [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor.
  Participants
    N0 | 18 | 20 | 38
    N1 | 7 | 8 | 15
    N2a | 3 | 2 | 5
    N2b | 19 | 19 | 38
    N2c | 15 | 13 | 28
    N3 | 2 | 1 | 3
Overall stage [Count of Participants; unit: Participants] — Overall cancer stage per American Joint Committee on Cancer (AJCC) 7th ed. combines tumor (T), regional lymph node (N), and distant metastasis (M) staging to determine an overall stage of II, III, or IV, ranging from least to most advanced, respectively. Stage II: T2/N0/M0; Stage III: T3/N0/M0 or T1-3/N1/M0; Stage IV: T4a/N0-1/M0 or T4b/any N/M0 or any T/N2-3/M0. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. The higher the number after the N, the greater the involvement of regional lymph nodes. M0 indicates no distant metastasis.
  Participants
    II | 1 | 0 | 1
    III | 18 | 20 | 38
    IV | 45 | 43 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive Without Progression (Progression-free Survival)
Description: An event for progression-free survival is local, regional, or distant disease progression or death due to any cause. Progression-free survival time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of survival times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided. Analysis occurred after 67 progressions or deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 7.1 years.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Number analyzed (Participants) | 64 | 63
percentage of participants | 34.6 [21.2 to 48.0] | 43.1 [30.1 to 56.1]
Statistical Analysis 1: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Hazard ratio (lapatinib/placebo) set at 0.65 (35% reduction), 1-sided alpha 0.20 (final test at 0.1803 accounting for 1 interim analysis), logrank test, 80% power, 69 events in 128 randomized (142 total enrolled) patients required. Final analysis at 67 (of 69) events drops power to 79%; Test type: Superiority; p = 0.3436, Log Rank; One-sided significance level = 0.1803; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.56 to 1.46] — Reference level = IMRT + cisplatin + placebo

2. Secondary Outcome: Percentage of Participants Alive (Overall Survival)
Description: An event for overall survival is death due to any cause. Overall survival time is defined as time from randomization to the date of death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of survival times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 7.1 years.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Number analyzed (Participants) | 64 | 63
percentage of participants | 55.1 [40.6 to 69.5] | 49.9 [35.5 to 64.3]
Statistical Analysis 1: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Superiority; p = 0.5836, Log Rank; One-sided significance level = 0.05; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.61 to 1.86] — Reference level = IMRT + cisplatin + placebo

3. Secondary Outcome: Percentage of Participants With Distant Metastases
Description: Failure for distant metastasis endpoint was defined as distant progression; local-regional failure and death due to any cause were considered competing risks. Distant metastasis time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Rates are estimated by the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 7.1 years.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Number analyzed (Participants) | 64 | 63
percentage of participants | 19.9 [10.1 to 32.2] | 12.4 [5.4 to 22.5]
Statistical Analysis 1: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Superiority; p = 0.1743, Log Rank; One-sided significance level = 0.05; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.25 to 1.65] — Reference level = IMRT + cisplatin + placebo

4. Secondary Outcome: Percentage of Participants With Treatment-related Grade 3 or Higher Adverse Events
Description: Adverse events (AE) were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to adverse event. "Treatment-related" is defined definitely, probably, or possibly related to treatment.
Time Frame: From start of treatment to last follow-up. Maximum follow-up at time of analysis was 7.1 years.
Population: Participants Who Started Protocol Treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Number analyzed (Participants) | 59 | 60
percentage of participants | 84.7 [73.0 to 92.8] | 86.7 [75.4 to 94.1]
Statistical Analysis 1: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Superiority; p = 0.7989, Fisher Exact; Two-sided significance level = 0.05

5. Secondary Outcome: Percentage of Participants Who Complied With Protocol Treatment
Description: Compliance with protocol treatment is defined as "per protocol" or "acceptable variation" per study chair review for IMRT, cisplatin, pre-IMRT lapatinib/placebo, concurrent lapatinib/placebo, and maintenance lapatinib/placebo. Rates of treatment compliance were compared between groups by a 2-sided Fisher's exact test.
Time Frame: From start of treatment to end of treatment (approximately 5 months from randomization).
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Number analyzed (Participants) | 64 | 63
percentage of participants
  IMRT | 76.6 [66.2 to 86.9] | 84.1 [75.1 to 93.2]
  Cisplatin | 90.6 [83.5 to 97.8] | 88.9 [81.1 to 96.6]
  Pre-IMRT lapatinib/placebo | 84.4 [75.5 to 93.3] | 87.3 [79.1 to 95.5]
  Concurrent lapatinib/placebo | 79.7 [69.8 to 89.5] | 84.1 [75.1 to 93.2]
  Maintenance lapatinib/placebo | 56.3 [44.1 to 68.4] | 49.2 [36.9 to 61.6]
Statistical Analysis 1: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Superiority; p = 0.3728, Fisher Exact — IMRT; Two-sided significance level = 0.05
Statistical Analysis 2: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Other; p = 0.7781, Fisher Exact — Cisplatin; Two-sided significance level = 0.05
Statistical Analysis 3: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Other; p = 0.8000, Fisher Exact — Pre-IMRT lapatinib/placebo; Two-sided significance level = 0.05
Statistical Analysis 4: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Other; p = 0.6459, Fisher Exact — Concurrent lapatinib/placebo; Two-sided significance level = 0.05
Statistical Analysis 5: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Other; p = 0.4792, Fisher Exact — Maintenance lapatinib/placebo; Two-sided significance level = 0.05

6. Secondary Outcome: Percentage of Participants With Local-regional Progression
Description: Failure for local-regional control endpoint was defined as local or regional progression, salvage surgery of the primary tumor with tumor present/unknown, salvage neck dissection with tumor present/unknown > 20 weeks after the end of radiation therapy, death due to study cancer without documented progression, or death due to unknown causes without documented progression; distant metastasis and death due to other causes were considered competing risks. Local-regional failure time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Failure rates are estimated by the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 7.1 years.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Number analyzed (Participants) | 64 | 63
percentage of participants | 33.7 [21.2 to 46.7] | 37.7 [25.0 to 50.4]
Statistical Analysis 1: Comparison: IMRT + Cisplatin + Placebo vs IMRT + Cisplatin + Lapatinib; Test type: Superiority; p = 0.6735, Log Rank; One-sided significance level = 0.05; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.62 to 2.17] — Reference level = IMRT + cisplatin + placebo

7. Secondary Outcome: Performance Status Scale for Head & Neck Cancer.
Time Frame: 3 months, 1 year, and 2 years
Reporting Status: Not Posted, anticipated posting 2023-09

8. Secondary Outcome: Functional Assessment of Cancer Therapy - Head & Neck.
Time Frame: 3 months, 1 year, and 2 years.
Reporting Status: Not Posted, anticipated posting 2023-09

9. Secondary Outcome: University of Michigan Xerostomia-Related Quality of Life Scale.
Time Frame: 3 months, 1 year, and 2 years.
Reporting Status: Not Posted, anticipated posting 2023-09

10. Secondary Outcome: HER2, EGFR, EMT as Biomarkers of Response.
Time Frame: End of Study
Population: No assays were performed, and no data were collected for this outcome measure. Specimen use will require funding separate from this trial.
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Weekly during radiation therapy, then every 3 months for years 1 and 2, every 6 months for years 3-5, then annually
Description: All-cause mortality was assessed in all randomized participants. Adverse events were assessed in participants who started protocol treatment
Arm/Group | IMRT + Cisplatin + Placebo | IMRT + Cisplatin + Lapatinib
All-Cause Mortality (participants affected / at risk) | 23/64 | 26/63
Serious Adverse Events (participants affected / at risk) | 26/59 | 31/60
Other Adverse Events (participants affected / at risk) | 59/59 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Cisplatin + Placebo (N=59) | IMRT + Cisplatin + Lapatinib (N=60)
Anemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 6 | 4
Esophagitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 7
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 6
Death NOS (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 0 | 2
Pain (General disorders) | 2 | 1
Sudden death NOS (General disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Injury to carotid artery (Injury, poisoning and procedural complications) | 1 | 0
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Creatinine increased (Investigations) | 2 | 2
Ejection fraction decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 8 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 8
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 4
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Cisplatin + Placebo (N=59) | IMRT + Cisplatin + Lapatinib (N=60)
Anemia (Blood and lymphatic system disorders) | 38 | 36
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 7 | 5
Sinus tachycardia (Cardiac disorders) | 4 | 1
Ear pain (Ear and labyrinth disorders) | 14 | 12
Hearing impaired (Ear and labyrinth disorders) | 18 | 15
Tinnitus (Ear and labyrinth disorders) | 23 | 14
Hyperthyroidism (Endocrine disorders) | 2 | 3
Hypothyroidism (Endocrine disorders) | 17 | 16
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 32 | 17
Dental caries (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 8 | 24
Dry mouth (Gastrointestinal disorders) | 47 | 46
Dyspepsia (Gastrointestinal disorders) | 8 | 8
Dysphagia (Gastrointestinal disorders) | 53 | 55
Esophageal pain (Gastrointestinal disorders) | 4 | 2
Esophageal stenosis (Gastrointestinal disorders) | 3 | 3
Esophagitis (Gastrointestinal disorders) | 3 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 5
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 12 | 18
Mucositis oral (Gastrointestinal disorders) | 45 | 48
Nausea (Gastrointestinal disorders) | 32 | 35
Oral pain (Gastrointestinal disorders) | 10 | 13
Salivary duct inflammation (Gastrointestinal disorders) | 5 | 6
Vomiting (Gastrointestinal disorders) | 20 | 25
Chills (General disorders) | 4 | 4
Edema face (General disorders) | 6 | 6
Edema limbs (General disorders) | 3 | 5
Fatigue (General disorders) | 49 | 49
Fever (General disorders) | 8 | 0
General disorders and administration site conditions - Other (General disorders) | 7 | 5
Localized edema (General disorders) | 4 | 8
Neck edema (General disorders) | 2 | 7
Non-cardiac chest pain (General disorders) | 4 | 6
Pain (General disorders) | 22 | 14
Infections and infestations - Other (Infections and infestations) | 5 | 4
Laryngitis (Infections and infestations) | 2 | 3
Lung infection (Infections and infestations) | 3 | 1
Mucosal infection (Infections and infestations) | 9 | 5
Skin infection (Infections and infestations) | 2 | 4
Upper respiratory infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 3 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 39 | 35
Fall (Injury, poisoning and procedural complications) | 2 | 4
Alanine aminotransferase increased (Investigations) | 12 | 14
Alkaline phosphatase increased (Investigations) | 9 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 7
Blood bilirubin increased (Investigations) | 4 | 10
CD4 lymphocytes decreased (Investigations) | 2 | 3
Creatinine increased (Investigations) | 18 | 19
Investigations - Other (Investigations) | 5 | 4
Lymphocyte count decreased (Investigations) | 22 | 26
Neutrophil count decreased (Investigations) | 22 | 13
Platelet count decreased (Investigations) | 16 | 14
Weight loss (Investigations) | 31 | 41
White blood cell decreased (Investigations) | 25 | 24
Anorexia (Metabolism and nutrition disorders) | 32 | 34
Dehydration (Metabolism and nutrition disorders) | 15 | 14
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 16 | 18
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 4
Hypernatremia (Metabolism and nutrition disorders) | 3 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 | 20
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 17 | 23
Hypomagnesemia (Metabolism and nutrition disorders) | 16 | 23
Hyponatremia (Metabolism and nutrition disorders) | 26 | 29
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 4
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 7 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 4 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 6
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 8 | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 12 | 17
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 5 | 2
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 9 | 6
Trismus (Musculoskeletal and connective tissue disorders) | 5 | 4
Dizziness (Nervous system disorders) | 5 | 8
Dysgeusia (Nervous system disorders) | 36 | 38
Headache (Nervous system disorders) | 13 | 12
Nervous system disorders - Other (Nervous system disorders) | 2 | 5
Neuralgia (Nervous system disorders) | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 11
Tremor (Nervous system disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 16 | 14
Confusion (Psychiatric disorders) | 4 | 1
Depression (Psychiatric disorders) | 10 | 11
Insomnia (Psychiatric disorders) | 13 | 20
Psychiatric disorders - Other (Psychiatric disorders) | 5 | 3
Acute kidney injury (Renal and urinary disorders) | 5 | 6
Hematuria (Renal and urinary disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 4 | 0
Urinary retention (Renal and urinary disorders) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 20
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 16
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 29 | 29
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 12 | 12
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Sore throat (Respiratory, thoracic and mediastinal disorders) | 21 | 25
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 7 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 7
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 | 4
Hot flashes (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 8 | 11
Hypotension (Vascular disorders) | 11 | 4
Lymphedema (Vascular disorders) | 6 | 6

LIMITATIONS AND CAVEATS:
A total of 69 progression-free survival (PFS) were required. As of September 13, 2020, the number of observed PFS events was 66. At the Radiation Therapy Oncology Group Foundation Data Monitoring Committee meeting on October 22, 2020, a decision was made to report the final results using data through November 30, 2020. This decision has a minor impact (<1%) on the power given that 67 PFS events are included in the final analysis of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT01711658/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT01711658/ICF_001.pdf